CLINICAL TRIAL: NCT05684354
Title: Validation of the Quality of Recovery-15 Score in Cardiac Surgery: The PROCARDS Study
Brief Title: Patient Reported Outcome (PRO) in CARDiac Surgery.
Acronym: PRO-CARDS
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC22_3088 PROCARDS
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Cardiac Surgery
Keywords: cardiac; surgery; postoperative care
MeSH Terms: interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient Reported Outcomes (PROs) — The day before or the morning before surgery, the patient filled the first QoR-15 scale alone or could be helped by one of the investigators in case of questions or difficulties.
  The second QoR-15 scale was distributed the day before or the day of discharge from the hospital

SUMMARY:
The use of Patient Reported Outcomes (PROs) in anaesthesia provides a measure of the patient's quality of postoperative recovery based on his/her own experience. The Quality-Of-Recovery-15 (QoR-15) is a widely used questionnaire which has never been validated in cardiac surgery patients.

This study aimed at validating the French version of the QoR-15 scale in a cohort of cardiac surgical patients. The QoR-15 scale would have similar psychometric properties and interpretability in assessing postoperative recovery in this population than in general surgery patients.

DETAILED DESCRIPTION:
The French version of the QoR-15 scale as validated by Demumieux et al was used in this study. Eligible patients were given oral and written information the day before or the morning before surgery. After patient agreed to participate, the first QoR-15 scale was distributed by one of the investigators. The patient filled in the questionnaire alone or could be helped by one of the investigators in case of questions or difficulties.

The second QoR-15 scale was distributed the day before or the day of discharge from the hospital and at the same time the patient was asked to rate his global recovery on a visual analog scale (VAS) graduated from 0 to 100 with 0 being the worst recovery and 100 the best recovery.

Patient demographic characteristics were collected including age, sex, body mass index (BMI), American Society of Anesthesiologists (ASA) physical status score, preoperative status of diabetes, hypertension, smoking status. Following perioperative data were recorded: type of surgery, duration of CPB, need for cardiac pacing or dobutamine support at the end of surgery, number of pleural and mediastinal chest tubes.

Postoperative complications were also recorded: surgical revision, atrial fibrillation requiring antiarrhythmic medication or anticoagulation, pulmonary oedema requiring depletion, drained pleural effusion, drained pneumothorax, radiological atelectasis, radiologic pneumonia, stroke with radiological diagnosis, sepsis as defined by Third International Consensus Definitions for Sepsis and Septic Shock [Sepsis-3], Heparin-induced thrombocytopenia (HIT) documented by Serotonin release assay test. Total dose of morphine used in ICU, length of stay (LOS) in ICU and hospital, duration of surgical drains and mortality at day 28 were also assessed.

Statistical analysis Sample size was The sample size was estimated at 150 patients and based on previous published studies(7,8) and guidelines recommending at least 10 subjects per item on the instrument scale(15). Data were reported as mean, median (inter-quartile range), or number (percentage) as appropriate. Correlations were calculated with Pearson correlation coefficient for Gaussian data or with Spearman correlation coefficient for non-Gaussian data. Factors associated with the QOR-15 score were searched by Analysis of Variance (ANOVA) for qualitative parameters and by linear regression for quantitative parameters. The null hypothesis was rejected if two-tailed P-value was inferior to 0.05

ELIGIBILITY:
Inclusion criteria:

* Patients over 18 years old
* Hospitalized for planned cardiac surgery among: coronary artery bypass grafting, valve plasty, valve replacement or ascending aortic surgery
* Patient not opposing his participation in the research

Non-inclusion criteria:

* Adults subject to legal protection (safeguard of justice, curatorship, guardianship)
* Persons deprived of liberty
* Patient unable to complete the questionnaire independently (cognitive deficit or patient who does not speak French)
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients scheduled for cardiac surgery under CPB including valve surgery, coronary artery bypass, ascending aorta surgery, combined procedure, and had given oral informed consent. Adults subject to legal protection (safeguard of justice, curatorship, guardianship), persons deprived of liberty, patients unable to complete the questionnaire independently (cognitive deficit or poor French comprehension) and pregnant or breastfeeding women were not included
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Assess the validity of QoR-15 in the post-operative period of cardiac surgery | Day 5
  Validity (the accuracy of a scale - does the QoR-15 measure what is intended: the quality of postoperative recovery). Convergent validity was tested by the hypothesis that there would be a positive correlation between the postoperative QoR-15 score and the global recovery assessment by the patient, or between the QoR-15 (postoperative-preoperative QoR-15 scores) and the global recovery assessment. Construct validity was tested by the hypothesis that there would be a negative association between the QoR-15 score and various known determinants of postoperative recovery

SECONDARY OUTCOMES:
Assess the Reliability of QoR-15 in the post-operative period of cardiac surgery | Day 5
  Reliability (the consistency of a scale) was tested by internal consistency (Cronbach's alpha)
Assess the Responsiveness of QoR-15 in the post-operative period of cardiac surgery | Day 5
  Responsiveness (ability of a scale to detect clinically important change) was assessed by Cohen size effect and standardized response mean.
Assess the Feasibility of QoR-15 in the post-operative period of cardiac surgery | Day 5
  Feasibility (applicability of a scale in practice) was evaluated by the successful completion rate

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire LE GAC, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided